CLINICAL TRIAL: NCT05784636
Title: Comparative Study on the Effectiveness, Comfort and Compliance of High-flow Nasal Oxygen Therapy and Noninvasive Mechanical Ventilation BiPAP Mode in the Treatment of Hypoxemia Patients
Brief Title: Comparative Study on the Effectiveness, Comfort and Compliance of HFNC and Noninvasive Mechanical Ventilation BiPAP Mode in the Treatment of Hypoxemia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2022039
Record Dates: First submitted 2022-09-19; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-11

CONDITIONS: Hypoxemia
Keywords: Hypoxemia, High-flow nasal cannula, Mechanical ventilation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive BiPAP ventilation treatment group (Experimental): Patients were first treated with HFNC on the basis of conventional treatment. The initial parameters were temperature: 31-37 °C, flow rate: 30-40 L/min, maintaining SpO2>92%, adjusting oxygen concentration according to blood oxygen saturation, and treatment duration was 24 h. After 24 h, patients were treated with non-invasive ventilator-assisted ventilation BiPAP mode until discharge
  Interventions: Device: Non-invasive BiPAP ventilation; Device: HFNC
- HFNC treatment group (Experimental): On the basis of conventional treatment, patients were first administered a noninvasive ventilator with the following initial parameters. BiPAP mode with an initial inspiratory pressure (IPAP) of 8-15 cmH2O and an initial expiratory pressure (EPAP) of 4-8 cmH2O. These parameters were adjusted according to the patient's specific conditions. After 24 hours of treatment, patients received HFNC until discharge.
  Interventions: Device: Non-invasive BiPAP ventilation; Device: HFNC

INTERVENTIONS:
Device: Non-invasive BiPAP ventilation — Patients were first treated with HFNC (High-flow nasal cannula) on the basis of conventional treatment. The initial parameters were temperature: 31-37 °C, flow rate: 30-40l /min, maintaining SpO2>92%, adjusting oxygen concentration according to blood oxygen saturation, and treatment duration was 24 h. After 24 h, patients were treated with non-invasive ventilator-assisted ventilation BiPAP mode until discharge.
  Other Names: HFNC
Device: HFNC — On the basis of conventional treatment, patients were first administered a noninvasive ventilator with the following initial parameters. BiPAP mode with an initial inspiratory pressure (IPAP) of 8-15 cmH2O and an initial expiratory pressure (EPAP) of 4-8 cmH2O. These parameters were adjusted according to the patient's specific conditions. After 24 hours of treatment, patients received HFNC (High-flow nasal cannula) until discharge.
  Other Names: Non-invasive BiPAP ventilation

SUMMARY:
Patients who met the inclusion criteria were included and signed an informed consent form, which complied with the requirements of the ethics committee of our unit. All subjects were inpatients. Subjects were randomized into two groups. patients in group A were first treated with HFNC on top of conventional treatment, and after 24 hours, patients were treated with non-invasive ventilator-assisted ventilation BiPAP mode until discharge. patients in group B were treated with a non-invasive ventilator on top of conventional treatment, and after 24 hours of treatment, patients were treated with HFNC until discharge. Patient information was collected during treatment.

DETAILED DESCRIPTION:
Patients who met the inclusion criteria were included and signed the informed consent, which met the requirements of the ethics committee of our unit. All subjects were hospitalized patients. Subjects were randomly divided into two groups. Patients in group A were treated with HFNC on the basis of conventional treatment. The initial parameters were: temperature:31-37℃, flow: 30-40l /min, SpO2 > 92% maintained, the oxygen concentration was adjusted according to the patient's oxygen saturation, and the treatment time was 24h. Twenty-four hours later, the patients were treated with non-invasive ventilator-assisted ventilation BiPAP mode until discharge. On the basis of conventional treatment, patients in group B were given a non-invasive ventilator with the following initial parameters: BiPaP mode, initial inspiratory pressure (IPAP) of 8-15cmH2O, initial expiratory pressure (EPAP) of 4-8cmH2O. The parameters were adjusted according to the specific conditions of the patients. After 24 hours of treatment, the patient was treated with HFNC until discharge. Patient information was collected during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. . PaO2 < 60mmHg, SpO2 < 92%(without oxygen inhalation);
2. Mild to moderate type I respiratory failure (100 mmHg < PaO/Fi02≤300 mmHg);

Exclusion Criteria:

1. Missing primary outcome measures
2. Terminal stage of various chronic diseases;
3. The patient or family members do not agree to NIV or HFNI treatment;
4. Severe type I respiratory failure (PaO2/Fi02≤100 mmHg)
5. Ventilation dysfunction (pH<7.30)
6. Contradictory breathing
7. The patient abandons or terminates treatment, automatically discharges or transfers to another hospital;
8. Serious diseases, such as organ function damage and sepsis;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
HR | At the time of enrollment in the clinical study
  Heart rate
HR | On the first hour after enrollment
  Heart rate
HR | On the second hour after enrollment
  Heart rate
HR | On the 6th hour after enrollment
  Heart rate
HR | On the 12th hour after enrollment
  Heart rate
HR | On the 24th hour after enrollment
  Heart rate
HR | On the 25th hour after enrollment (On the first hour after crossover)
  Heart rate
HR | On the 26th hour after enrollment (On the second hour after crossover)
  Heart rate
HR | On the 30th hour after enrollment (On the 6th hour after crossover)
  Heart rate
HR | On the 36th hour after enrollment (On the 12th hour after crossover)
  Heart rate
HR | On the 48th hour after enrollment (On the 24th hour after crossover)
  Heart rate
HR | On the third day after enrollment (On the 48th hour after crossover)
  Heart rate
HR | On the 4th day after enrollment (On the third day after crossover)
  Heart rate
HR | On the 5th day after enrollment (On the 4th day after crossover)
  Heart rate
HR | On the 6th day after enrollment (On the 5th day after crossover)
  Heart rate
HR | On the 7th day after enrollment (On the 6th day after crossover)
  Heart rate
HR | On the 8th day after enrollment (On the 7th day after crossover)
  Heart rate
HR | On the 9th day after enrollment (On the 8th day after crossover)
  Heart rate
RR | At the time of enrollment in the clinical study
  Respiratory rate
RR | On the first hour after enrollment
  Respiratory rate
RR | On the second hour after enrollment
  Respiratory rate
RR | On the 6th hour after enrollment
  Respiratory rate
RR | On the 12th hour after enrollment
  Respiratory rate
RR | On the 24th hour after enrollment
  Respiratory rate
RR | On the 25th hour after enrollment (On the first hour after crossover)
  Respiratory rate
RR | On the 26th hour after enrollment (On the second hour after crossover)
  Respiratory rate
RR | On the 30th hour after enrollment (On the 6th hour after crossover)
  Respiratory rate
RR | On the 36th hour after enrollment (On the 12th hour after crossover)
  Respiratory rate
RR | On the 48th hour after enrollment (On the 24th hour after crossover)
  Respiratory rate
RR | On the third day after enrollment (On the 48th hour after crossover)
  Respiratory rate
RR | On the 4th day after enrollment (On the third day after crossover)
  Respiratory rate
RR | On the 5th day after enrollment (On the 4th day after crossover)
  Respiratory rate
RR | On the 6th day after enrollment (On the 5th day after crossover)
  Respiratory rate
RR | On the 7th day after enrollment (On the 6th day after crossover)
  Respiratory rate
RR | On the 8th day after enrollment (On the 7th day after crossover)
  Respiratory rate
RR | On the 9th day after enrollment (On the 8th day after crossover)
  Respiratory rate
BP | At the time of enrollment in the clinical study
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the first hour after enrollment
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the second hour after enrollment
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 6th hour after enrollment
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 12th hour after enrollment
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 24th hour after enrollment
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 25th hour after enrollment (On the first hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 26th hour after enrollment (On the second hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 30th hour after enrollment (On the 6th hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 36th hour after enrollment (On the 12th hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 48th hour after enrollment (On the 24th hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the third day after enrollment (On the 48th hour after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 4th day after enrollment (On the third day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 5th day after enrollment (On the 4th day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 6th day after enrollment (On the 5th day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 7th day after enrollment (On the 6th day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 8th day after enrollment (On the 7th day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
BP | On the 9th day after enrollment (On the 8th day after crossover)
  Blood pressure (Includes systolic and diastolic blood pressure)
SO2 | At the time of enrollment in the clinical study
  Pulse oxygen saturation
SO2 | On the first hour after enrollment
  Pulse oxygen saturation
SO2 | On the second hour after enrollment
  Pulse oxygen saturation
SO2 | On the 6th hour after enrollment
  Pulse oxygen saturation
SO2 | On the 12th hour after enrollment
  Pulse oxygen saturation
SO2 | On the 24th hour after enrollment
  Pulse oxygen saturation
SO2 | On the 25th hour after enrollment (On the first hour after crossover)
  Pulse oxygen saturation
SO2 | On the 26th hour after enrollment (On the second hour after crossover)
  Pulse oxygen saturation
SO2 | On the 30th hour after enrollment (On the 6th hour after crossover)
  Pulse oxygen saturation
SO2 | On the 36th hour after enrollment (On the 12th hour after crossover)
  Pulse oxygen saturation
SO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  Pulse oxygen saturation
SO2 | On the third day after enrollment (On the 48th hour after crossover)
  Pulse oxygen saturation
SO2 | On the 4th day after enrollment (On the third day after crossover)
  Pulse oxygen saturation
SO2 | On the 5th day after enrollment (On the 4th day after crossover)
  Pulse oxygen saturation
SO2 | On the 6th day after enrollment (On the 5th day after crossover)
  Pulse oxygen saturation
SO2 | On the 7th day after enrollment (On the 6th day after crossover)
  Pulse oxygen saturation
SO2 | On the 8th day after enrollment (On the 7th day after crossover)
  Pulse oxygen saturation
SO2 | On the 9th day after enrollment (On the 8th day after crossover)
  Pulse oxygen saturation
pH | At the time of enrollment in the clinical study
  Degree of pH in arterial blood
pH | On the 24th hour after enrollment
  Degree of pH in arterial blood
pH | On the 48th hour after enrollment (On the 24th hour after crossover)
  Degree of pH in arterial blood
pH | On the third day after enrollment (On the 48th hour after crossover)
  Degree of pH in arterial blood
pH | On the 4th day after enrollment (On the 3th day after crossover)
  Degree of pH in arterial blood
pH | On the 5th day after enrollment (On the 4th day after crossover)
  Degree of pH in arterial blood
pH | On the 6th day after enrollment (On the 5th day after crossover)
  Degree of pH in arterial blood
pH | On the 7th day after enrollment (On the 6th day after crossover)
  Degree of pH in arterial blood
pH | On the 8th day after enrollment (On the 7th day after crossover)
  Degree of pH in arterial blood
pH | On the 9th day after enrollment (On the 8th day after crossover)
  Degree of pH in arterial blood
PaO2 | At the time of enrollment in the clinical study
  Partial arterial oxygen pressure
PaO2 | On the 24th hour after enrollment
  Partial arterial oxygen pressure
PaO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  Partial arterial oxygen pressure
PaO2 | On the third day after enrollment (On the 48th hour after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 4th day after enrollment (On the 3th day after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 5th day after enrollment (On the 4th day after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 6th day after enrollment (On the 5th day after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 7th day after enrollment (On the 6th day after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 8th day after enrollment (On the 7th day after crossover)
  Partial arterial oxygen pressure
PaO2 | On the 9th day after enrollment (On the 8th day after crossover)
  Partial arterial oxygen pressure
SaO2 | At the time of enrollment in the clinical study
  Arterial oxygen saturation
SaO2 | On the 24th hour after enrollment
  Arterial oxygen saturation
SaO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial oxygen saturation
SaO2 | On the third day after enrollment (On the 48th hour after crossover)
  Arterial oxygen saturation
SaO2 | On the 4th day after enrollment (On the third day after crossover)
  Arterial oxygen saturation
SaO2 | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial oxygen saturation
SaO2 | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial oxygen saturation
SaO2 | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial oxygen saturation
SaO2 | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial oxygen saturation
SaO2 | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial oxygen saturation
PCO2 | At the time of enrollment in the clinical study
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 24th hour after enrollment
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the third day after enrollment (On the 48th hour after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 4th day after enrollment (On the third day after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 5th day after enrollment (On the 4th day after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 6th day after enrollment (On the 5th day after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 7th day after enrollment (On the 6th day after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 8th day after enrollment (On the 7th day after crossover)
  partial pressure of carbon dioxide in arterial blood
PCO2 | On the 9th day after enrollment (On the 8th day after crossover)
  partial pressure of carbon dioxide in arterial blood
FiO2 | At the time of enrollment in the clinical study
  Fraction of inspiration O2
FiO2 | On the 24th hour after enrollment
  Fraction of inspiration O2
FiO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  Fraction of inspiration O2
FiO2 | On the third day after enrollment (On the 48th hour after crossover)
  Fraction of inspiration O2
FiO2 | On the 4th day after enrollment (On the third day after crossover)
  Fraction of inspiration O2
FiO2 | On the 5th day after enrollment (On the 4th day after crossover)
  Fraction of inspiration O2
FiO2 | On the 6th day after enrollment (On the 5th day after crossover)
  Fraction of inspiration O2
FiO2 | On the 7th day after enrollment (On the 6th day after crossover)
  Fraction of inspiration O2
FiO2 | On the 8th day after enrollment (On the 7th day after crossover)
  Fraction of inspiration O2
FiO2 | On the 9th day after enrollment (On the 8th day after crossover)
  Fraction of inspiration O2
Lac | At the time of enrollment in the clinical study
  Lactic acid in arterial blood
Lac | On the 24th hour after enrollment
  Lactic acid in arterial blood
Lac | On the 48th hour after enrollment (On the 24th hour after crossover)
  Lactic acid in arterial blood
Lac | On the third day after enrollment (On the 48th hour after crossover)
  Lactic acid in arterial blood
Lac | On the 4th day after enrollment (On the third day after crossover)
  Lactic acid in arterial blood
Lac | On the 5th day after enrollment (On the 4th day after crossover)
  Lactic acid in arterial blood
Lac | On the 6th day after enrollment (On the 5th day after crossover)
  Lactic acid in arterial blood
Lac | On the 7th day after enrollment (On the 6th day after crossover)
  Lactic acid in arterial blood
Lac | On the 8th day after enrollment (On the 7th day after crossover)
  Lactic acid in arterial blood
Lac | On the 9th day after enrollment (On the 8th day after crossover)
  Lactic acid in arterial blood
Glu | At the time of enrollment in the clinical study
  Arterial blood glucose in arterial blood
Glu | On the 24th hour after enrollment
  Arterial blood glucose in arterial blood
Glu | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial blood glucose in arterial blood
Glu | On the third day after enrollment (On the 48th hour after crossover)
  Arterial blood glucose in arterial blood
GLu | On the 4th day after enrollment (On the third day after crossover)
  Arterial blood glucose in arterial blood
Glu | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial blood glucose in arterial blood
Glu | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial blood glucose in arterial blood
Glu | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial blood glucose in arterial blood
Glu | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial blood glucose in arterial blood
Glu | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial blood glucose in arterial blood
A-aDO2 | At the time of enrollment in the clinical study
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 24th hour after enrollment
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the third day after enrollment (On the 48th hour after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 4th day after enrollment (On the third day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 5th day after enrollment (On the 4th day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 6th day after enrollment (On the 5th day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 7th day after enrollment (On the 6th day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 8th day after enrollment (On the 7th day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
A-aDO2 | On the 9th day after enrollment (On the 8th day after crossover)
  The difference between the oxygen partial pressure of alveolar air and the oxygen partial pressure of arterial blood
BE | At the time of enrollment in the clinical study
  Base excess in arterial blood
BE | On the 24th hour after enrollment
  Base excess in arterial blood
BE | On the 48th hour after enrollment (On the 24th hour after crossover)
  Base excess in arterial blood
BE | On the third day after enrollment (On the 48th hour after crossover)
  Base excess in arterial blood
BE | On the 4th day after enrollment (On the third day after crossover)
  Base excess in arterial blood
BE | On the 5th day after enrollment (On the 4th day after crossover)
  Base excess in arterial blood
BE | On the 6th day after enrollment (On the 5th day after crossover)
  Base excess in arterial blood
BE | On the 7th day after enrollment (On the 6th day after crossover)
  Base excess in arterial blood
BE | On the 8th day after enrollment (On the 7th day after crossover)
  Base excess in arterial blood
BE | On the 9th day after enrollment (On the 8th day after crossover)
  Base excess in arterial blood
RI | At the time of enrollment in the clinical study
  Respiratory Index
RI | On the 24th hour after enrollment
  Respiratory Index
RI | On the 48th hour after enrollment (On the 24th hour after crossover)
  Respiratory Index
RI | On the third day after enrollment (On the 48th hour after crossover)
  Respiratory Index
RI | On the 4th day after enrollment (On the third day after crossover)
  Respiratory Index
RI | On the 5th day after enrollment (On the 4th day after crossover)
  Respiratory Index
RI | On the 6th day after enrollment (On the 5th day after crossover)
  Respiratory Index
RI | On the 7th day after enrollment (On the 6th day after crossover)
  Respiratory Index
RI | On the 8th day after enrollment (On the 7th day after crossover)
  Respiratory Index
RI | On the 9th day after enrollment (On the 8th day after crossover)
  Respiratory Index
Arterial blood HCO3- concentration | At the time of enrollment in the clinical study
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 24th hour after enrollment
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the third day after enrollment (On the 48th hour after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 4th day after enrollment (On the third day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood HCO3- concentration | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial blood HCO3- concentration，including arterial blood HCO3- std concentration
Arterial blood K+ concentration | At the time of enrollment in the clinical study
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 24th hour after enrollment
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the third day after enrollment (On the 48th hour after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 4th day after enrollment (On the third day after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial blood K+ concentration
Arterial blood K+ concentration | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial blood K+ concentration
Arterial blood Ca2+ concentration | At the time of enrollment in the clinical study
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 24th hour after enrollment
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the third day after enrollment (On the 48th hour after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 4th day after enrollment (On the third day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Ca2+ concentration | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial blood Ca2+ concentration
Arterial blood Na+ concentration | At the time of enrollment in the clinical study
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 24th hour after enrollment
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 48th hour after enrollment (On the 24th hour after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the third day after enrollment (On the 48th hour after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 4th day after enrollment (On the third day after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 5th day after enrollment (On the 4th day after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 6th day after enrollment (On the 5th day after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 7th day after enrollment (On the 6th day after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 8th day after enrollment (On the 7th day after crossover)
  Arterial blood Na+ concentration
Arterial blood Na+ concentration | On the 9th day after enrollment (On the 8th day after crossover)
  Arterial blood Na+ concentration
TCO2 | At the time of enrollment in the clinical study
  Total carbon dioxide in arterial blood
TCO2 | On the 24th hour after enrollment
  Total carbon dioxide in arterial blood
TCO2 | On the 48th hour after enrollment (On the 24th hour after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the third day after enrollment (On the 48th hour after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 4th day after enrollment (On the third day after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 5th day after enrollment (On the 4th day after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 6th day after enrollment (On the 5th day after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 7th day after enrollment (On the 6th day after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 8th day after enrollment (On the 7th day after crossover)
  Total carbon dioxide in arterial blood
TCO2 | On the 9th day after enrollment (On the 8th day after crossover)
  Total carbon dioxide in arterial blood
HCT | At the time of enrollment in the clinical study
  hematocrit in arterial blood
HCT | On the 24th hour after enrollment
  hematocrit in arterial blood
HCT | On the 48th hour after enrollment (On the 24th hour after crossover)
  hematocrit in arterial blood
HCT | On the third day after enrollment (On the 48th hour after crossover)
  hematocrit in arterial blood
HCT | On the 4th day after enrollment (On the third day after crossover)
  hematocrit in arterial blood
HCT | On the 5th day after enrollment (On the 4th day after crossover)
  hematocrit in arterial blood
HCT | On the 6th day after enrollment (On the 5th day after crossover)
  hematocrit in arterial blood
HCT | On the 7th day after enrollment (On the 6th day after crossover)
  hematocrit in arterial blood
HCT | On the 8th day after enrollment (On the 7th day after crossover)
  hematocrit in arterial blood
HCT | On the 9th day after enrollment (On the 8th day after crossover)
  hematocrit in arterial blood
tHbc | At the time of enrollment in the clinical study
  Total hemoglobin in arterial blood
tHbc | On the 24th hour after enrollment
  Total hemoglobin in arterial blood
tHbc | On the 48th hour after enrollment (On the 24th hour after crossover)
  Total hemoglobin in arterial blood
tHbc | On the third day after enrollment (On the 48th hour after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 4th day after enrollment (On the third day after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 5th day after enrollment (On the 4th day after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 6th day after enrollment (On the 5th day after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 7th day after enrollment (On the 6th day after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 8th day after enrollment (On the 7th day after crossover)
  Total hemoglobin in arterial blood
tHbc | On the 9th day after enrollment (On the 8th day after crossover)
  Total hemoglobin in arterial blood
height | At the time of enrollment in the clinical study
  m
Weight | At the time of enrollment in the clinical study
  Kg
gender | At the time of enrollment in the clinical study
  Male and female
age | At the time of enrollment in the clinical study
  year
WBC | On the first day after enrollment
  The number of white blood cells in venous blood
WBC | up to 9 days
  The number of white blood cells in venous blood
NEU | On the first day after enrollment
  The number of Neutrophil granulocyte in venous blood
NEU | up to 9 days
  The number of Neutrophil granulocyte in venous blood
LYM | On the first day after enrollment
  The number of Venous blood lymphocytes in venous blood
LYM | up to 9 days
  The number of Venous blood lymphocytes in venous blood
EOS | On the first day after enrollment
  The number of Venous blood eosinophils in venous blood
EOS | up to 9 days
  The number of Venous blood eosinophils in venous blood
BAS | On the first day after enrollment
  The number of Venous blood Basophils in venous blood
BAS | up to 9 days
  The number of Venous blood Basophils in venous blood
MON | On the first day after enrollment
  The number of Venous blood Monocyte cell in venous blood
MON | up to 9 days
  The number of Venous blood Monocyte cell in venous blood
RBC | On the first day after enrollment
  The number of red blood cells in venous blood
RBC | up to 9 days
  The number of red blood cells in venous blood
HGB | On the first day after enrollment
  The number of haemoglobin in venous blood
HGB | up to 9 days
  The number of haemoglobin in venous blood
HCT | On the first day after enrollment
  hematocrit in venous blood
HCT | up to 9 days
  hematocrit in venous blood
MCV | On the first day after enrollment
  Mean Corpuscular Volume in venous blood
MCV | up to 9 days
  Mean Corpuscular Volume in venous blood
MCH | On the first day after enrollment
  Mean Corpuscular Haemoglobin Concentration in venous blood
MCH | up to 9 days
  Mean Corpuscular Haemoglobin Concentration in venous blood
RDW | On the first day after enrollment
  red blood cell distribution width in venous blood
RDW | up to 9 days
  red blood cell distribution width in venous blood
PLT | On the first day after enrollment
  platelet in venous blood
PLT | up to 9 days
  platelet in venous blood
PDW | On the first day after enrollment
  Platelet distributionwidth in venous blood
PDW | up to 9 days
  Platelet distributionwidth in venous blood
MPV | On the first day after enrollment
  Mean Platelet Volume in venous blood
MPV | up to 9 days
  Mean Platelet Volume in venous blood
plateletcrit | On the first day after enrollment
  plateletcrit in venous blood
plateletcrit | up to 9 days
  plateletcrit in venous blood
CRP | On the first day after enrollment
  C-reactive protein in venous blood
CRP | up to 9 days
  C-reactive protein in venous blood
PCT | On the first day after enrollment
  Procalcitonin in venous blood
PCT | up to 9 days
  Procalcitonin in venous blood
NT-proBNP | On the first day after enrollment
  NT-proBNP in venous blood
NT-proBNP | up to 9 days
  NT-proBNP in venous blood
ESR | On the first day after enrollment
  erythrocytesedimentationrate in venous blood
ESR | up to 9 days
  erythrocytesedimentationrate in venous blood
PT | On the first day after enrollment
  prothrombin time in venous blood
PT | up to 9 days
  prothrombin time in venous blood
APTT | On the first day after enrollment
  activated partial thromboplastin time in venous blood
APTT | up to 9 days
  activated partial thromboplastin time in venous blood
TT | On the first day after enrollment
  Thrombin time in venous blood
TT | up to 9 days
  Thrombin time in venous blood
D-Di | On the first day after enrollment
  D-Dimer in venous blood
D-Di | up to 9 days
  D-Dimer in venous blood
ALT | On the first day after enrollment
  alanine transaminase in venous blood
ALT | up to 9 days
  alanine transaminase in venous blood
AST | On the first day after enrollment
  Aspartate Transaminase in venous blood
AST | up to 9 days
  Aspartate Transaminase in venous blood
PA | On the first day after enrollment
  Serum prealbumin in venous blood
PA | up to 9 days
  Serum prealbumin in venous blood
TP | On the first day after enrollment
  Total serum protein in venous blood
TP | up to 9 days
  Total serum protein in venous blood
ALB | On the first day after enrollment
  Albumin protein in venous blood
ALB | up to 9 days
  Albumin protein in venous blood
GLB | On the first day after enrollment
  Globulin globulin in venous blood
GLB | up to 9 days
  Globulin globulin in venous blood
Cr | On the first day after enrollment
  creatinine in venous blood
Cr | up to 9 days
  creatinine in venous blood
BUN | On the first day after enrollment
  Urea nitrogen in venous blood
BUN | up to 9 days
  Urea nitrogen in venous blood
Cys-C | On the first day after enrollment
  Cystatin C in venous blood
Cys-C | up to 9 days
  Cystatin C in venous blood
eGFR | On the first day after enrollment
  Estimate glomerular filtration rate in venous blood
eGFR | up to 9 days
  Estimate glomerular filtration rate in venous blood
Respiratory support time | during hospitalization, approximately 9 days
  Daily respiratory support time after patients were enrolled in the clinical study，h/Day
Relief time for dyspnea | during hospitalization, approximately 9 days
  Remission time of dyspnea after intervention
Tracheal intubation | during hospitalization, approximately 9 days
  Yes or No
Stay in the ICU | during hospitalization, approximately 9 days
  Yes or No
Complications | during hospitalization, approximately 9 days
  Facial injury, flatulence，Gastroesophageal reflux，Dry throat, sore throat，pneumothorax，Eye irritation discomfort，Low blood pressure.
Outcome of disease | during hospitalization, approximately 9 days
  Get better, get worse, die
Total bilirubin | On the first day after enrollment
  Serum total bilirubin in venous blood
Total bilirubin | up to 9 days
  Serum total bilirubin in venous blood
DBIL | On the first day after enrollment
  Direct bilirubin in venous blood
DBIL | up to 9 days
  Direct bilirubin in venous blood
IBIL | On the first day after enrollment
  Indirect bilirubin in venous blood
IBIL | up to 9 days
  Indirect bilirubin in venous blood
Diaphragm mobility | At the time of enrollment in the clinical study
  The patient is lying in a flat position. The convex array probe is placed at the junction of the anterior axillary line, midclavicular line, and rib margin (bilaterally), with the probe mark facing outward and downward for measurement.
Diaphragm mobility | On the 24th hour after enrollment
  The patient is lying in a flat position. The convex array probe is placed at the junction of the anterior axillary line, midclavicular line, and rib margin (bilaterally), with the probe mark facing outward and downward for measurement.
Diaphragm mobility | On the 48th hour after enrollment (On the 24th hour after crossover)
  The patient is lying in a flat position. The convex array probe is placed at the junction of the anterior axillary line, midclavicular line, and rib margin (bilaterally), with the probe mark facing outward and downward for measurement.
Diaphragm mobility | up to 9 days
  The patient is lying in a flat position. The convex array probe is placed at the junction of the anterior axillary line, midclavicular line, and rib margin (bilaterally), with the probe mark facing outward and downward for measurement.
Diaphragm thickness | At the time of enrollment in the clinical study
  Includes end-inspiratory diaphragm thickness and end-expiratory diaphragm thickness；The patient is lying flat on the bed. A linear array probe is placed in the mid-axillary line or between the anterior and mid-axillary lines between the eighth and tenth ribs, and measurements are taken.
Diaphragm thickness | On the 24th hour after enrollment
  Includes end-inspiratory diaphragm thickness and end-expiratory diaphragm thickness；The patient is lying flat on the bed. A linear array probe is placed in the mid-axillary line or between the anterior and mid-axillary lines between the eighth and tenth ribs, and measurements are taken.
Diaphragm thickness | On the 48th hour after enrollment (On the 24th hour after crossover)
  Includes end-inspiratory diaphragm thickness and end-expiratory diaphragm thickness；The patient is lying flat on the bed. A linear array probe is placed in the mid-axillary line or between the anterior and mid-axillary lines between the eighth and tenth ribs, and measurements are taken.
Diaphragm thickness | up to 9 days
  Includes end-inspiratory diaphragm thickness and end-expiratory diaphragm thickness；The patient is lying flat on the bed. A linear array probe is placed in the mid-axillary line or between the anterior and mid-axillary lines between the eighth and tenth ribs, and measurements are taken.

SECONDARY OUTCOMES:
Patient compliance to the treatment | during hospitalization, approximately 9 days
  Patients were managed for compliance with the treatment.Dependent judgment
  1. Complete dependence: patients actively cooperate with medical staff in treatment
  2. Partial dependence: in most cases, patients can cooperate with the treatment, and in a few cases, patients resist the treatment but receive treatment after being enlightened by the medical staff.
  3. Non-dependence: patients have strong resistance and resistance, so that they are unable to use ventilators or nasal high-flow humidification instruments.
Kolcaba Comfort Scale (GCQ) assessment assesses patient comfort | during hospitalization, approximately 9 days
  Kolcaba's General Comfort Questionnaire (GCQ) is composed of 28 items from 4 dimensions: physiological, psychological, spiritual, socio-cultural and environmental. The modification Scale adopts 1 to 4Likert Scale, with 1 indicating strongly disagree and 4 indicating strongly agree. In the negative question, 1 means strongly agree and 4 means strongly disagree. A higher score indicates more comfort.
Dyspnea rating scale | during hospitalization, approximately 9 days
  According to the degree of dyspnea and symptoms of the patient, the lowest score is 0, the highest score is 10.

CONTACTS AND LOCATIONS:
Overall Officials: Dedong Ma, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Milesi C, Essouri S, Pouyau R, Liet JM, Afanetti M, Portefaix A, Baleine J, Durand S, Combes C, Douillard A, Cambonie G; Groupe Francophone de Reanimation et d'Urgences Pediatriques (GFRUP). High flow nasal cannula (HFNC) versus nasal continuous positive airway pressure (nCPAP) for the initial respiratory management of acute viral bronchiolitis in young infants: a multicenter randomized controlled trial (TRAMONTANE study). Intensive Care Med. 2017 Feb;43(2):209-216. doi: 10.1007/s00134-016-4617-8. Epub 2017 Jan 26. PMID 28124736
- [Result] Lewis SR, Baker PE, Parker R, Smith AF. High-flow nasal cannulae for respiratory support in adult intensive care patients. Cochrane Database Syst Rev. 2021 Mar 4;3(3):CD010172. doi: 10.1002/14651858.CD010172.pub3. PMID 33661521
- [Result] Chen BX, Ou Q, Pan MX. [A cross-sectional survey of treatment acceptance and influence factors in patients with obstructive sleep apnea]. Zhonghua Yi Xue Za Zhi. 2018 May 29;98(20):1578-1581. doi: 10.3760/cma.j.issn.0376-2491.2018.20.010. Chinese. PMID 29886648